CLINICAL TRIAL: NCT02868047
Title: Establishing Standards for Normal Pancreatic EUS
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Timothy Gardner, Associate Profesor, Department of Medicine, Dartmouth-Hitchcock Medical Center
Other Study IDs: 21516
Record Dates: First submitted 2014-01-02; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Pancreatitis
Keywords: chronic pancreatitis; endoscopic ultrasound
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Suspected Chronic Pancreatitis: Included patients will be those scheduled for an upper endoscopic ultrasound examination with suspected chronic pancreatitis
  Interventions: Procedure: Endoscopic Ultrasound
- NOT Suspected Chronic Pancreatitis: Included patients will be those scheduled for an upper endoscopic ultrasound examination without suspected chronic pancreatitis.
  Interventions: Procedure: Endoscopic Ultrasound

INTERVENTIONS:
Procedure: Endoscopic Ultrasound — Patients will undergo elective upper endoscopic ultrasound to evaluate the pancreas in patients both with and without chronic pancreatitis

SUMMARY:
There is tremendous variability in regard to provider perception of findings on EUS for chronic pancreatitis. This study performs tandem EUS exams between expert endosonogrpahers to determine the validity of minimal standard criteria.

DETAILED DESCRIPTION:
Chronic pancreatitis is a very challenging disease to diagnose as their is no gold standard for diagnosis. Increasingly, endoscopic ultrasound (EUS) has been used as a means of diagnosing chronic pancreatitis. However, there are questions about whether intra-rater reliability and/or validity are high enough to warrant using EUS to make the diagnosis of chronic pancreatitis.

The purpose of this observational study is to determine the degree of correlation between two expert endosonographers in evaluating minimal standard criteria (MST) in the same patient during the same EUS exam. Patients both with and without chronic pancreatitis will be included in the study to try and determine the validity and reliability of back-to-back EUS examinations.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing upper EUS for evaluation of the pancreas

Exclusion Criteria:

* pregnancy
* age less than 18
* inability to provide written informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include patients who are scheduled for an elective EUS for evaluation of their pancreas. Patients will be those with and without suspected chronic pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Hyperechoic Strands | Day 1
Number of Patients with Hyperechoic Foci | Day 1
Number of Patients with Lobular Contour | Day 1
Number of Patients with Cysts | Day 1
Number of Patients with Duct Irregularity | Day 1
Number of Patients with Ductal Calculi | Day 1
Number of Patients with Hyperechoic Duct Wall | Day 1
Number of Patients with Dilated Dilated Side Branches | Day 1
Number of Patients with Dilated Pancreatic Duct | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No